CLINICAL TRIAL: NCT05309889
Title: A Prospective Observational Study of Clinical Efficacy, Complications, and Prognosis in Patients With Sepsis in ICU
Brief Title: A Prospective Observational Study of Sepsis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSEC-KY-KS-2022-009
Record Dates: First submitted 2022-03-30; First posted 2022-04-04 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-03

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- high exposure level: Patients have a high level of exposure factors
  Interventions: Other: no intervention
- low exposure level: Patients have a low level of exposure factors
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Sepsis is a life-threatening organ dysfunction caused by a dysregulated host response to infection and is associated with high morbidity and mortality. Sepsis3 gives sepsis a broad definition, reflecting the heterogeneity of the disease. So we need a precise treatment with a stratification of patient prognosis in order to reduce mortality in patients with sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who met the Sepsis3 diagnostic criteria.

Exclusion Criteria:

* Absence of laboratory test items (blood routine examination, coagulation function, liver function, biochemistry, urine routine examination, urine renal function, urine protein, etc.) >20%.
* Admission in ICU less than 48 hours.
* Patient with psychiatric disorders.
* Under 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were hospitalized in the ICU of Sun Yat-sen Memorial Hospital of Sun Yat-sen University and met the Sepsis 3 diagnostic criteria.
Sampling Method: Non-Probability Sample
Enrollment: 174 (Estimated)
Dates: Start 2022-05-12 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
mortality rate | 28 days after diagnosis of sepsis
  all-cause deaths that occurred in 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guangzhou, China